CLINICAL TRIAL: NCT01430039
Title: Syndecan-1 as a Surrogate Marker for Inflammatory Bowel Disease
Brief Title: Syndecan-1 a Surrogate Marker for IBD
Acronym: syndecan1
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 03.09.11.01; 31.08.11 (Registry Identifier: syndecan-1 and inflammatory bowel disease)
Record Dates: First submitted 2011-08-28; First posted 2011-09-07 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2012-03

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Crohn's disease; ulcerative colitis; Syndecan-1
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Blood Specimen Collection; Syndecan-1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Venous blood sample for syndecan-1 levels, blood count, CRP levels,serum albumin and total protein
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Crohn's, ulcerative colitis: Patients with diagnosed with Crohn's disease or ulcerative colitis who agreed to participate in the study and singed informed consent and answered a Crohn's disease activity index questioner for Crohn's disease or the ulcerative colitis activity index questioner for ulcerative colitis.
  Interventions: Procedure: Blood sample - venous blood 10 ml.
- No disease: Healthy subjects with no known inflammatory disease. For basal serum levels of syndecan 1
  Interventions: Procedure: blood sample

INTERVENTIONS:
Procedure: blood sample — Blood sample from a peripheral vein, 10ml total for blood count, total serum : protein, albumin, LDH, C-reactive protein,syndecan-1
  Other Names: Syndecan-1
  Groups: No disease
Procedure: Blood sample - venous blood 10 ml. — venous blood sample from a peripheral vein, 10ml total for blood count, total serum : protein, albumin, LDH, C-reactive protein,syndecan-1
  Other Names: Syndecan-1
  Groups: Crohn's, ulcerative colitis

SUMMARY:
Syndecan-1 is a protein on the surface intestinal cells. previous studies proved low levels of mucosal syndecan-1 levels on the surface of intestinal cells is patients with acute and chronic inflammation due to inflammatory bowel disease.

this protein might shed from cell surface to the serum. The investigators wish to prove that elevated serum levels of syndecan-1 may be predictive of disease presence, extent and severity, that buy taking a simple blood sample from patients diagnosed with inflammatory bowel disease and comparing to normal subjects and to other markers.

DETAILED DESCRIPTION:
One of the main hypothesis for the etiology of Inflammatory bowel disease (IBD) is an inappropriate and ongoing activation of the mucosal immune system in response to the presence of normal luminal flora. This aberrant response is most likely facilitated by defects in both the barrier function and the mucosal immune system of the intestinal epithelium. Syndecans are a class proteoglycans that take part in both cell adhesion and growth factor binding. Of the four known syndecan core proteins, syndecan-1 (CD138) and one of the best studied of this group and is also the relevant to the this study as it is expressed on the basolateral surface of columnar epithelial cells of the colon. Syndecan-1 functions as an integral membrane protein that participates in cell proliferation, cell migration and cell matrix interactions in the GI tract. Evidence for a reduction of syndecan-1 expression in the regenerating epithelium that overlies inflamed tissue was reported in both acute and chronic inflammation. This protein that is lost from the inflamed mucosal membrane might shed to the serum. Elevated serum levels of syndecan-1 may be predictive of disease presence and extent.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* no other concurrent inflammatory disease
* formal diagnosis of inflammatory bowel disease i.e Crohn's disease, Ulcerative colitis

Exclusion Criteria:

* pregnancy
* fever at time of sample taking

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Normal population, having no known inflammatory disease
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2011-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Elevated serum syndecan-1 levels as a bio marker for IBD | one year
  elevated serum syndecan-1 levels in patients with IBD compared to control

SECONDARY OUTCOMES:
Serum syndecan-1 levels and disease severity Crohn's | one year
  Relationship between clinical data CDAI in crohn's patients and serum syndecan-1 levels
Serum syndecan-1 levels and disease severity ulcerative colitis | one year
  Relationship between clinical data UCAI ulcerative colitis patients and serum syndecan-1 levels
Serum syndecan-1 levels and C reactive protein(CRP) Crohn's | one year
  Relationship between lab data CRP levels in crohn's patients and serum syndecan-1 levels
Serum syndecan-1 levels and C reactive protein(CRP) ulcerative colitis | one year
  Relationship between serum CRP levels and serum syndecan-1 levels in patients with ulcerative colitis

CONTACTS AND LOCATIONS:
Overall Officials: Assaf Stein, Md, Principal Investigator — resident
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

REFERENCES:
- [Background] Yablecovitch D, Shabat-Simon M, Aharoni R, Eilam R, Brenner O, Arnon R. Beneficial effect of glatiramer acetate treatment on syndecan-1 expression in dextran sodium sulfate colitis. J Pharmacol Exp Ther. 2011 May;337(2):391-9. doi: 10.1124/jpet.110.174276. Epub 2011 Feb 10. PMID 21310817
- [Background] Bartlett AH, Hayashida K, Park PW. Molecular and cellular mechanisms of syndecans in tissue injury and inflammation. Mol Cells. 2007 Oct 31;24(2):153-66. PMID 17978567
- [Background] Bode L, Salvestrini C, Park PW, Li JP, Esko JD, Yamaguchi Y, Murch S, Freeze HH. Heparan sulfate and syndecan-1 are essential in maintaining murine and human intestinal epithelial barrier function. J Clin Invest. 2008 Jan;118(1):229-38. doi: 10.1172/JCI32335. PMID 18064305
- [Background] Carey DJ. Syndecans: multifunctional cell-surface co-receptors. Biochem J. 1997 Oct 1;327 ( Pt 1)(Pt 1):1-16. doi: 10.1042/bj3270001. PMID 9355727
- [Background] Seidel C, Sundan A, Hjorth M, Turesson I, Dahl IM, Abildgaard N, Waage A, Borset M. Serum syndecan-1: a new independent prognostic marker in multiple myeloma. Blood. 2000 Jan 15;95(2):388-92. PMID 10627439
- [Background] Principi M, Day R, Marangi S, Burattini O, De Francesco V, Ingrosso M, Pisani A, Panella C, Forbes A, Di Leo A, Francavilla A, Ierardi E. Differential immunohistochemical expression of syndecan-1 and tumor necrosis factor alpha in colonic mucosa of patients with Crohn's disease. Immunopharmacol Immunotoxicol. 2006;28(2):185-95. doi: 10.1080/08923970600815048. PMID 16873088
- [Background] Gotte M. Syndecans in inflammation. FASEB J. 2003 Apr;17(6):575-91. doi: 10.1096/fj.02-0739rev. PMID 12665470
- [Background] Gaffney PR, O'Leary JJ, Doyle CT, Gaffney A, Hogan J, Smew F, Annis P. Response to heparin in patients with ulcerative colitis. Lancet. 1991 Jan 26;337(8735):238-9. doi: 10.1016/0140-6736(91)92201-c. No abstract available. PMID 1670865
- [Background] Day RM, Mitchell TJ, Knight SC, Forbes A. Regulation of epithelial syndecan-1 expression by inflammatory cytokines. Cytokine. 2003 Mar 7;21(5):224-33. doi: 10.1016/s1043-4666(03)00091-7. PMID 12824007
- [Background] Day R, Ilyas M, Daszak P, Talbot I, Forbes A. Expression of syndecan-1 in inflammatory bowel disease and a possible mechanism of heparin therapy. Dig Dis Sci. 1999 Dec;44(12):2508-15. doi: 10.1023/a:1026647308089. PMID 10630505